CLINICAL TRIAL: NCT03378908
Title: Medical Nutrition Therapy in Gestational Diabetes Mellitus: Comparison of Different Number of Meals. A Pilot Study
Brief Title: Carbohydrates Distribution in Pregnancy Study
Acronym: CHiPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Hospital Arnau de Vilanova (Other); Institut de Recerca Biomèdica de Lleida (Other); Universitat de Lleida (Other); Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Principal Investigator, Didac Mauricio, Head of Endocrinology and Nutrition, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DMG-0001
Record Dates: First submitted 2017-12-04; First posted 2017-12-20 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: medical therapy nutrition; meal; carbohydrates; intervention; food intake
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Masking Description: Glycemic profile will be collected with a blind-sensor during the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment 6 meals (No Intervention): Diet will be distributed with 6 meals (breakfast, lunch, dinner and 3 snacks). This is the usual diet prescribed for women with GDM at the Department of Endocrinology and Nutrition of both Centers. Energy intake distribution: 25% breakfast, 5% snack, 30% lunch, 10% snack, 25% dinner and 5% snack.
- Intervention Treatment 3 meals (Experimental): Diet will be distributed in 3 meals (breakfast, lunch and dinner). Each meal will consist of the addition of the conventional meal and the next snack. Energy intake will be distributed: 30% breakfast (25% breakfast + 5% snack), 40% lunch (30% lunch + 10% snack) and 30% dinner (25% dinner and 5% snack).
  Interventions: Behavioral: Intervention Treatment

INTERVENTIONS:
Behavioral: Intervention Treatment — Both groups (conventional and treatment) will have the same nutritional composition, with 40% carbohydrates, 20% protein and 40% total fat (preferently monounsaturated fatty acids).
  Arms: Intervention Treatment 3 meals

SUMMARY:
Hypothesis: Patients with Gestational Diabetes Mellitus (GDM) have a high risk to develop complications during pregnancy, puerperium and in the newborn. At present there are not scientific evidences about the optimal distribution of meals in the medical nutrition therapy (MNT) and their relationship with glycemic control.

Aim: To explore and compare ketonemia and glycemic profile in patients with GDM that follow a MNT distributed in 6 or 3 meals. Besides, we want to explore the differences between both treatments in glucose dynamics.

Methods: The study design is a randomized, crossover and multicentric trial. A sample of 10 patients with GDM will be recruited in the Department of Endocrinology and Nutrition from both centres. In a randomized manner patients will follow the conventional treatment (a carbohydrate-controlled diet distributed in 6 meals: 3 main meals and 3 snacks) and the intervention treatment (a carbohydrate-controlled diet distributed in 3 meals: breakfast, lunch and dinner). They will be randomized to begin with one of the two treatments, and after two weeks they will be switched to the other treatment. Patients will wear a blinded continuous glucose monitoring device (iPro2-TM, Medtronic) during the entire study period.

Inclusion criteria:

* Women with GDM diagnosed in 24-28 weeks.
* Age 18-40 years.
* Pregnancy age of 28-32 weeks.
* Caucasian.
* Body mass index ≤ 35 Kg/m2.

Exclusion criteria:

* Unability to understand the dietary recommendations and/or to perform self-management of glycemia, ketonuria or ketonemia.
* A low adherence to MNT.
* Problems with written and/or oral communication.
* Presence of comorbidities other than obesity, hypertension and dyslipidemia.
* Insulin-need criteria within 3 first days of the beginning of the study (fasting glucose ≥90mg/dL, postprandial glucose 1-hour ≥140mg/dL).

Clinical and sociodemographic variables will be assessed. Dietary records and blood samples will be collected. Daily basal ketonuria and ketonemia before each meal will be assessed. Glycemic profile will be collected with a blind-sensor during the four weeks of the intervention study. Generalized linear model analysis will be performed. Statistical power will be 80% and significance level will be set at 0.05. Written informed consent will be collected from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Women with GDM diagnosed in 24-28 weeks.
* Age 18-40 years.
* Pregnancy age of 28-32 weeks.
* Caucasian.
* Body mass index ≤ 35Kg/m2.
* Firs-time mother.

Exclusion Criteria:

* Disability to understand the dietary recommendations and/or to perform self-management of glycemia, ketonuria or ketonemia.
* A low adherence to MNT.
* Problems with write and oral communication.
* Other comorbidities differed of obesity, hypertension and dyslipidemia.
* Insulin criteria within 3 first days of study (fasting glucose ≥90mg/dL, postprandial glucose 1-hour ≥140mg/dL).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Preprandial ketonemia | 4 weeks (2 weeks with the conventional treatment and 2 weeks with the intervention treatment)
  Before the 3 main meals every day.
Glycemic profile below pregnancy target capillary blood glucose concentration | 4 weeks (2 weeks with conventional treatment and 2 weeks with intervention treatment)
  Self monitoring blood glucose levels: pre meals < 90 mg/dL, 1 hour post meals <140mg/dL

SECONDARY OUTCOMES:
Area under the curve of interstitial glucose levels | Time Frame: 4 weeks (2 weeks with conventional treatment and 2 weeks with intervention treatment)
  Blinded continuous glucose monitoring data, iPro2, Medtronic (r)): diurnal (from 7 am to 11 pm) and nocturnal (from 11pm to 7 am)
Fetal Macrosomia | Through study completion, 4 weeks
  US assessed fetal weight, adjusted for national standardized charts
Newborn body weight adjusted for gestational age (national standardized charts) | At delivery
  Large for gestational age > 90th centile, small for gestational age < 10th centile
Newborn hypoglycemia | 48 hours from delivery
  Serum glycemia <40 mg/dL in the first 48 hours of life
Postpartum glucose tolerance of the mother | 6 weeks after delivery
  Plasma glucose levels fasting and 120 minutes after a 75 g oral glucose load
Point-of-care glycated hemoglobin (HbA1c) | Every 2 weeks from the date of randomization until the last visit of the study
  DCA Vantage Analyzer, Siemens ®

CONTACTS AND LOCATIONS:
Overall Officials: Didac Mauricio, MD PHD, Study Director — Germans Trias i Pujol Hospital
Locations (2):
- Spain (2):
  - Berta Soldevila, Badalona, Barcelona
  - Marta Hernández, Lleida